CLINICAL TRIAL: NCT04220749
Title: A Phase II Randomized Trial for HPV-Negative Oropharyngeal Squamous Cell Carcinoma: Radiotherapy vs. Trans-Oral Surgery (ORATOR)
Brief Title: Radiotherapy vs. Trans-Oral Surgery for HPV-Negative Oropharyngeal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORATOR 3
Record Dates: First submitted 2020-01-06; First posted 2020-01-07 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Head and Neck Cancer; Oropharyngeal Squamous Cell Carcinoma
Keywords: Radiotherapy; Trans-Oral Surgery; HPV-Negative; Randomized
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiation; Drug Therapy; Neck Dissection

STUDY DESIGN:
Intervention Model Description: 2 Arm study randomized in a 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1, Radiation +/- Chemotherapy (Active Comparator): Standard Treatment (Radiation +/- Chemotherapy)
  Interventions: Radiation: Radiation
- Arm 2, TOS + Neck Dissection (Experimental): Trans-oral Surgery (TOS) + Neck Dissection (plus radiation is required)
  Interventions: Procedure: Trans-Oral Surgery (TOS) + Neck Dissection

INTERVENTIONS:
Radiation: Radiation — Standard of Care: Radiation +/- Chemotherapy
  Other Names: Chemotherapy, if required
  Arms: Arm 1, Radiation +/- Chemotherapy
Procedure: Trans-Oral Surgery (TOS) + Neck Dissection — Trans-Oral Surgery (TOS) + Neck Dissection (plus radiation, if required)
  Other Names: Radiation, if required
  Arms: Arm 2, TOS + Neck Dissection

SUMMARY:
The goal of this randomized phase II study is a formal comparison of radiotherapy versus trans-oral surgery as the primary treatment of HPV-negative patients with early-stage oropharyngeal carcinoma.

DETAILED DESCRIPTION:
This study is designed as a randomized phase II study. Patients will be randomized between current standard of care treatment (Arm 1) vs. TOS (Arm 2) in a 1:1 ratio. Additionally, patients will be stratified according to T stage (T1 vs. T2); N stage (N0/1 vs. N2/3)

The randomized phase II design is required for three reasons:

1. The randomization will provide an appropriate control group to serve as a comparator for the experimental arm. Historical or contemporaneous non-randomized controls would not be appropriate due to the multitude of biases that could be introduced by patient selection and other confounders.
2. A small sample size will allow for adequate power to assess for progression-free survival, and also an assessment of quality of life, overall survival and toxicity.
3. The results will allow for a decision as to whether a multi-institutional phase III trial is warranted, and inform the design of such a trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Willing to provide informed consent
* ECOG performance status 0-2
* Histologically confirmed squamous cell carcinoma
* HPV-negative tumor, as determined by: negative p16 status, real time PCR or in-situ hybridization. Central confirmation is not required prior to randomization. Equivocal/uncertain HPV status will be allowed on trial.
* Primary tumor site in the oropharynx (includes tonsil, soft palate, base of tongue, walls of oropharynx)
* Tumor stage: T1 or T2, with likely negative resection margins at surgery
* Nodal stage: N0-3. Patients with positive nodal disease and extranodal extension on imaging may be included at the surgeon's discretion, if the nodal disease is deemed resectable by the operating surgeon.
* Eligible for curative intent treatment, with likely negative resection margins at surgery. For patients where adequate transoral access is in question, they will first undergo an examination under anesthesia prior to randomization to ensure adequate exposure can be obtained.
* Blood work obtained within 4 weeks prior to randomization, with adequate bone marrow function, hepatic, and renal function, as determined by the investigator.
* Patient assessed by a radiation oncologist and surgeon and presented at multidisciplinary tumor board prior to randomization. If not feasible, case can be discussed with study Principal Investigator.

Exclusion Criteria:

* Serious medical comorbidities or other contraindications to radiotherapy, chemotherapy or surgery
* Prior history of head and neck cancer within 5 years
* Prior head and neck radiation at any time
* Metastatic disease
* Inability to attend full course of radiotherapy or follow-up visits
* Prior invasive malignant disease unless disease-free for at least 5 years or more, with the exception of non-melanoma skin cancer
* Unable or unwilling to complete QOL questionnaires
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Disease-Specific Survival | 5 years
  Time from randomization to death from cancer

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Time from randomization to death from any cause
Progression-Free Survival | 5 years
  Defined as time from randomization to death from any cause
Local-Regional Failure | 5 years
  Defined as time from randomization to first local-regional failure (analyzed as cumulative incidence function with death as competing event)
Distant Failure | 5 years
  Defined as time from randomization to first distant failure or metastasis (analyzed as cumulative incidence function with death as competing event)
Any Failure | 5 years
  Defined as time from randomization to first local-regional failure or distant failure, whichever occurs first (analyzed as cumulative incidence function with death as competing event)
Quality of Life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: MD Anderson Dysphagia Inventory (MDADI)
Quality of Life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: EORTC QLQ-C30
Quality of Life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: H&N35 scale
Quality of Life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: Voice Handicap Index (VHI-10)
Quality of Life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: Neck Dissection Impairment Index (NDII)
Quality of Life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: Patient Neurotoxicity Questionnaire (PNQ)
Toxicity profile of both study arms using the National Cancer Institute Common Toxicity Criteria (NCI-CTC) Version 4 | Randomization until 5 years follow up
  To determine toxicity profile of both study arms using the National Cancer Institute Common Toxicity Criteria (NCI-CTC) Version 4
Feeding tube rate at 1 year | Baseline to 1 year post treatment
  Measure other functional measurements such as feeding tube rate at 1 year
CTCAE Dysphagia Grade | Baseline to 5 years post treatment
  Measure other functional measurements such as CTCAE Dysphagia grade

CONTACTS AND LOCATIONS:
Overall Officials: Danielle MacNeil, M.D., Principal Investigator — London Regional Cancer Program, London Health Sciences Centre
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada